CLINICAL TRIAL: NCT02342899
Title: Medium Cost Effectiveness of Automated Non-Invasive Ventilation Outpatient Set Up vs Standard Fixed Level Non-Invasive Ventilation Inpatient Set Up In Obese Patients With Chronic Respiratory Failure
Brief Title: Cost Effectiveness of Outpatient Set-up of Automated NIV in Obese Patients With Chronic Respiratory Failure
Acronym: OPIP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Guy's and St Thomas' NHS Foundation Trust (Other)
Collaborators: Philips Electronics Nederland B.V. acting through Philips CTO organization (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 139750
Record Dates: First submitted 2015-01-13; First posted 2015-01-21 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Obesity Hypoventilation Syndrome; Chronic Respiratory Failure
MeSH Terms: conditions — Obesity Hypoventilation Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Goup (Active Comparator): Inpatient initiation of noninvasive ventilation.
  Interventions: Device: Inpatient NIV Set Up using spontaneous/timed (S/T) mode pressure support ventilation (Manufactured by Philips-Respironics)
- Intervention Group (Active Comparator): Initiated on NIV during an elective outpatient clinic review during which an arterial blood gas measurement will be obtained to confirm the presence of chronic respiratory failure.
  Interventions: Device: Outpatient NIV Set Up using AVAPS AE (Manufactured by Philips-Respironics)

INTERVENTIONS:
Device: Outpatient NIV Set Up using AVAPS AE (Manufactured by Philips-Respironics) — Intervention set ups will follow a standard protocol for the automated device (A40 AVAPS-AE machine;Manufactured by Philips-Respironics, Murraysville, Pittsburgh, US) and patients will be discharged with the machine and a full face mask or nasal interface. Patients will then undergo a 1-2 night home oximetry study to ensure adequate control of overnight oxygenation. Patients will be reviewed clinically as an outpatient at 6 weeks and adherence to non-invasive ventilation will be evaluated and an arterial blood gas measurement will be undertaken. A full clinical review and optimisation of NIV and interface will be performed at this visit. Patients will be reviewed at 3 months as an inpatient where overnight transcutaneous carbon dioxide level and SpO2 studies will be performed. All other patient-centred, physician-centred and healthcare utilisation measurements will be assessed at baseline, 6 weeks and 3 months.
  Arms: Intervention Group
Device: Inpatient NIV Set Up using spontaneous/timed (S/T) mode pressure support ventilation (Manufactured by Philips-Respironics) — The patient will follow a specialist nurse-led protocolised set up of spontaneous/timed (S/T) mode pressure support ventilation (A40 AVAPS-AE machine; Manufactured by Philips-Respironics, Murraysville, Pittsburgh, US) using limited respiratory polygraphy, including overnight TcCO2 (Trascutaneous Carbon Dioxide) and SpO2 (Oxygen Saturation) studies. Following the inpatient set-up, patients will be reviewed as an outpatient at 6 weeks and adherence with non-invasive ventilation will be evaluated and arterial blood gas measurements will be performed. Patients will then be reviewed at 3 months as an inpatient where overnight respiratory polygraphy, TcCO2 and SpO2 studies will be repeated. All other patient-centred, physician-centred measurements and healthcare utilisation measurements will be assessed at baseline, 6 weeks and 3 months.
  Arms: Control Goup

SUMMARY:
Obesity is an escalating issue, with an accompanying increase in referrals of patients with obesity-related respiratory failure. Currently, these patients are electively admitted to hospital for initiation of non-invasive ventilation (NIV), but it is unknown whether outpatient initiation is as effective as inpatient set-up. The investigators hypothesise that outpatient set up using an auto-titrating NIV device will be more cost effective than nurse-led inpatient titration and set-up.

The investigators will undertake a multi-national, multi-centre randomised controlled trial.

Subjects will be randomised to receiving usual inpatient set-up, which will include nurse-led initiation of NIV or outpatient set-up with an automated NIV device. Subjects will be stratified according to trial site, gender and previous use of NIV or continuous positive airway pressure. Assuming 10% drop out rate, a total sample of 82 patients will be required. Cost effectiveness will be evaluated using standard treatment costs and health service utilisation and using health related quality of life measures (SRI and EQ5D). Change in the severe respiratory insufficiency (SRI) questionnaire will be based on analysis of covariance (ANCOVA) adjusting for the baseline measurements between the two arms of patients.

DETAILED DESCRIPTION:
There is an increase of patients with hypercapnic respiratory failure as a consequence of obesity. The current treatment options for patients with obesity related respiratory failure is non-invasive ventilation (NIV). This has shown to reduce partial pressure of arterial carbon dioxide (PaCO2) and improves symptoms such as dyspnea (breathlessness)and enhances quality of life. NIV has also shown to increase physical activity (using actigraphy)and there can be associated weight reduction after three months of initiation.

Currently, the length of an inpatient stay for NIV set up is between 4.5 and 6 days. As yet it is unknown whether or not a patient can be set up onto NIV as effectively on an outpatient basis using an AE-AVAPS (Automatic Expiratory Positive Airway Pressure - Average Volume Assured Pressure Support) algorithm compared to the usual practice of inpatient titration by specialist respiratory nurses. Furthermore, the cost effectiveness of outpatient initiation vs inpatient initiation is unknown in this group of patients.

This will be the first trial to assess the cost effectiveness of such a set up.

ELIGIBILITY:
Inclusion Criteria:

* Obese patients with chronic respiratory failure
* Age > 18 years
* Chronic hypercapnia (daytime PaCO2 > 6.0kPa)
* Evidence of sleep disordered breathing on overnight oximetry study (4% oxygen desaturation index >10events per hour and/or >30% of the total analysis time with an SpO2 < 90%)
* Patients with a recent acute episode requiring non-invasive ventilation will need a minimum of 2 weeks stability prior to enrolment into the trial (no NIV requirement for 2 weeks and pH (Inverse logarithm of hydrogen ion concentration) ≥ 7.3)
* BMI ≥ 35kg/m2
* FEV1/FVC (Forced Expiratory Volume at 1 second/Forced Vital Capacity) > 70%

Exclusion Criteria:

* Persistent hypercapnic respiratory acidosis defined as pH <7.30
* Severe hypoxic and/or hypercapnic respiratory failure defined as a PaO2 (Partial Pressure of Oxygen)< 7.0kPa and/or a PaCO2 > 9kPa (kilopascal)
* Failure to tolerate NIV during initiation or if required to treat acute decompensation
* Hypercapnic respiratory failure requiring intubation within the last 28 days
* Hypercapnic respiratory failure secondary to an identifiable cause other than obesity
* Acute coronary syndrome or unstable angina
* Cognitive impairment that would prevent informed consent into the trial and/or inability to comply with the protocol
* Psychiatric disease necessitating anti-psychotic medication, ongoing treatment for drug or alcohol addiction, persons of no fixed abode post-discharge
* Patients undergoing renal replacement therapy
* Patients with co-existent cancer and a prognosis likely to be less than 12-months
* Critical peripheral vascular disease awaiting re-vascularisation procedure (or claudication distance <100 metres)
* Stroke with hemiparesis
* Age <18 years
* Pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2015-03-01 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Medium Term Cost-Effectiveness | 3 months
  To evaluate the medium term cost effectiveness of outpatient non-invasive ventilation set-up with an automated device compared with inpatient nurse-led protocolised fixed level non-invasive ventilation set-up in obese patients with chronic respiratory failure at 3 months

SECONDARY OUTCOMES:
Health Related Quality of Life | 3 months
  To evaluate the health related quality of life improvements between outpatient non-invasive ventilation set-up and inpatient set-up at 3 months
Gas Exchange Improvements | 3 months
  To evaluate the gas exchange improvements between outpatient non-invasive ventilation set-up and inpatient set-up at 3 months.

CONTACTS AND LOCATIONS:
Overall Officials: Nick Hart, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (6):
- France (2):
  - Hôpital Universitaire, de Grenoble, Grenoble
  - Rouen University Hospital, Rouen
- United Kingdom (4):
  - Leeds Teaching Hospital NHS Foundation Trust, Leeds, Yorkshire
  - Royal Free Hospital, London
  - Guys and St Thomas NHS Foundation, London
  - Royal Brompton and Harefield NHS Foundation Trust, London

IPD SHARING:
Plan to Share IPD: No
No plan to share individual participant data

REFERENCES:
- [Derived] Murphy PB, Patout M, Arbane G, Mandal S, Kaltsakas G, Polkey MI, Elliott M, Muir JF, Douiri A, Parkin D, Janssens JP, Pepin JL, Cuvelier A, Flach C, Hart N. Cost-effectiveness of outpatient versus inpatient non-invasive ventilation setup in obesity hypoventilation syndrome: the OPIP trial. Thorax. 2023 Jan;78(1):24-31. doi: 10.1136/thorax-2021-218497. Epub 2022 Sep 2. PMID 36342884